CLINICAL TRIAL: NCT00486304
Title: Phase I Randomized, Double-blind, Placebo-controlled Trial of the Effect of Temporary Dietary Antioxidant Depletion on Tumor Growth and Cachexia in Head and Neck Cancer Patients Receiving Chemoradiation Therapy
Brief Title: Low Antioxidant Diet in Controlling Cachexia in Patients With Oropharyngeal Cancer Receiving Chemotherapy and Radiation Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LCCC 0523; CDR0000549772 (Other: PDQ number)
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Cachexia; Head and Neck Cancer; Weight Changes
Keywords: cachexia; weight changes; recurrent oropharyngeal cancer; stage I oropharyngeal cancer; stage II oropharyngeal cancer; stage III oropharyngeal cancer; stage IV oropharyngeal cancer
MeSH Terms: conditions — Cachexia; Head and Neck Neoplasms; Body Weight Changes; Oropharyngeal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antioxidant-deficient diet (ADD) (Experimental)
  Interventions: Other: ADD
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: ADD — The ADD has a composition of 65% carbohydrate, 20% fat, and 15% protein. The diet will be completely depleted of vitamins A, E and beta-carotene; it will have 10 mg of vitamin C (6.5% of RDA) added per person per day
  Arms: Antioxidant-deficient diet (ADD)
Other: Placebo — Jevity 1.5 (1.5 cal/mL) will be used for the placebo patients in this study. This will simulate the standard of care for patients not on the ADD. Jevity 1.5 is an isotonic, fiber-fortified, high-nitrogen liquid formula providing complete, balanced nutrition for patients requiring short- or long-term tube feeding, given once per day
  Arms: Placebo

SUMMARY:
RATIONALE: Eating a diet that is low in antioxidants may control cachexia in patients with oropharyngeal cancer.

PURPOSE: This randomized phase I trial is studying the side effects of a low antioxidant diet in controlling cachexia in patients with oropharyngeal cancer receiving chemotherapy and radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of the antioxidant-deficient diet (ADD) in controlling cachexia in patients with oropharyngeal cancer receiving chemoradiotherapy.

Secondary

* Determine the safety of the ADD as measured by quality of life, peripheral DNA damage, and change in body weight.
* Determine the effectiveness of the ADD on tumor growth and surrogate markers of tumor growth.
* Determine whether the ADD is effective in improving the tumor cachexia syndrome in these patients.
* Determine whether there is a serum metabolomic signature for the ADD.

OUTLINE: This a prospective, randomized, double-blind, placebo-controlled study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients consume a standard diet 3 times a day for 8 weeks.
* Arm II: Patients consume an antioxidant-deficient diet (ADD) 3 times a day for 8 weeks. Patients receive replacement vitamins in week 9.

All patients receive planned chemoradiotherapy in weeks 3-8.

Quality of life, body composition (by dual-energy x-ray absorptiometry), weight, and resting energy expenditure (by indirect calorimetry) are assessed at baseline and at week 8.

Blood samples are collected at baseline and at 8 weeks. Samples are evaluated for cytokine levels; evidence of DNA damage from peripheral blood lymphocytes; and serum signature characteristic to ADD by multinuclear MRI spectroscopy. Patients undergo a tumor biopsy in week 4 for research studies. Samples are collected and evaluated for generation of reactive oxygen species by using antibodies against oxidatively modified DNA and lipids; apoptosis using TdT-mediated dUTP nick-end labeling assay and classical morphological criteria; and levels of the tumor toxohormones lipid mobilizing factor and proteolysis inducing factor by real time-PCR, northern blotting, and western blotting methods.

After completion of study therapy, patients are followed once during weeks 9-12.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy-proven carcinoma of the oropharynx (regardless of primary diagnosis or recurrence)
* No active treatment for disease within the past 4 weeks

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Feeding tubes allowed
* Prior malignancies allowed provided all of the following criteria are met:

  * Patient has undergone potentially curative therapy for all prior malignancies
  * There has been no evidence of any prior malignancies within the past 5 years (except for successfully treated cervical or non-melanoma skin cancer with no evidence of recurrences)
  * Patient is deemed by their treating physician to be at low risk for recurrence from prior malignancies
* Must be able to speak English
* Must have adequate home refrigeration
* No intractable vomiting
* No ascites or clinical/ultrasound evidence of fluid retention
* No uncontrolled hypertension
* No severe congestive heart failure
* No pneumonia
* No severe infections
* No known HIV positivity
* No coexisting medical condition that would preclude study compliance
* No decisionally-impaired individuals
* No history of abetalipoproteinemia (Bassen-Kornzweig syndrome)
* No history of spinocerebellar ataxia
* No history of chronic cholestatic hepatobiliary disease
* No history of diagnosed vitamin E deficiency
* No history of protein-energy malnutrition (marasmus or kwashiorkor)
* No history of disorders related to malabsorption (e.g., celiac disease, sprue, cystic fibrosis, duodenal bypass, congenital partial obstruction of the jejunum, obstruction of the bile ducts, giardiasis, or cirrhosis)
* No history of achlorhydria

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-02; Primary Completion 2007-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Number of people with adverse events | 70 days
  Estimate the safety of the antioxidant-deficient diet (ADD) by measuring the frequency of grade 3 or 4 adverse events, per CTCAE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Marion Couch, MD, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States